CLINICAL TRIAL: NCT03557944
Title: Team Approach to Polypharmacy Evaluation and Reduction Pharmacy
Brief Title: Team Approach to Polypharmacy Evaluation and Reduction (Pharmacy)
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: McMaster University (Other)
Collaborators: Canadian Institutes of Health Research (CIHR) (Other Government); David Braley and Nancy Gordon Chair in Family Medicine (Other); RxISK (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 4619
Record Dates: First submitted 2018-06-05; First posted 2018-06-15 (Actual); Last update posted 2023-03-15 (Actual); Status verified 2023-03

CONDITIONS: Multi-morbidity; Medication Therapy Management; Polypharmacy

STUDY DESIGN:
Intervention Model Description: Single-arm, longitudinal cohort feasibility study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- TAPER (Experimental): The intervention is medication reduction. This arm is comprised of:
  1. Medication reconciliation
  2. Identification of patient priorities for care
  3. Identification of medications that are potentially appropriate for discontinuation/dose reduction
  4. Linked pharmacist/family physician consultations with patient to discuss medication with intention to reduce
  5. Identification of medications for trial of discontinuation/dose reduction (shared decision making)
  6. Pause of medication and clinical monitoring
  Interventions: Other: Medication reduction

INTERVENTIONS:
Other: Medication reduction — Systematic approach to reduction in polypharmacy.
  Other Names: Medication discontinuation/dose reduction

SUMMARY:
In an aging population, most seniors suffer from multiple chronic conditions. When the number of medications taken is ≥5 (polypharmacy), the burden of taking multiple concurrent medications can do more harm than good. Seniors take an average of 7 regular medications and studies link polypharmacy with adverse effects on morbidity, function and health service use. However, it is not clear to what extent these are reversible if medication burden is reduced.

This trial will test the effects on medication numbers and patient health outcomes of an intervention to polypharmacy. This study will test a program focused on medication reduction number and dose. Prioritizing medications according to the patient's preference as reducing the dose also reduces the risk of drug side effects.

Patients, aged 70 years of age or older and taking ≥5 medications will receive the TAPER program. The program involves information gathering from the patient, including systematically seeking patients priorities and preferences, medication review with the pharmacist and then a consultation with the family doctor. The intervention is focused on discontinuing/reducing the dose of medications where possible using a 'pause and monitor' framework to assess the need for restart. An electronic program that detects drug adverse effects and flags potentially inappropriate medications will be integrated into an electronic clinical pathway incorporating monitoring and follow-up systems.

This study will examine whether implementing a deprescribing care pathway with community pharmacists as point-of-entry can signal improvements in prescribing and patient health outcomes in older adults with polypharmacy.

DETAILED DESCRIPTION:
This study uses a single-arm, longitudinal cohort feasibility design. Patients will receive the intervention following baseline data collection. Initial baseline data collection from the patient will include information on demographics, medications, and illness characteristics. The patient will then attend an appointment with a pharmacist to review medications appropriate for discontinuation/dose reduction, after which the patient will meet with their family physician to discuss patient preferences for discontinuation/dose reduction. Both health care providers will have access to TaperMD, a web-based program linked to evidence and tools to support reduction in polypharmacy. Follow-up research assessments will take place at one week, 3 months and 6 months (study end). Outcome assessments and a semi-structured interview will take place at the 6 month appointment.

ELIGIBILITY:
Inclusion Criteria:

* Aged 70 years of age or older
* Patient must have a family doctor
* Participating family doctor as most responsible provider
* Currently taking 5 or more long-term medications
* Has not had a recent comprehensive medication review
* Patient willing to try discontinuation

Exclusion Criteria:

* English language or cognitive skills inadequate to understand and respond to rating scales
* Terminal illness or other circumstance precluding 6 month study period

Min Age: 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2019-06-16 (Actual); Primary Completion 2023-10 (Estimated); Study Completion 2024-06 (Estimated)

PRIMARY OUTCOMES:
Feasibility (recruitment number) | 6 months
  Number of people who are invited to participate in the study.

SECONDARY OUTCOMES:
Feasibility (proportion consented) | 6 months
  Number of participants who consent divided by the number of potential participants invited.
Feasibility (proportion completed) | 6 months
  Number of participants who complete 6-month data collection divided by the number of people who consented.
Feasibility (barriers to recruitment) | 6 months
  Challenges to recruitment as identified by pharmacists via field notes and interviews.
Feasibility (time to complete surveys) | Baseline, 6 months
  Total time to complete all surveys
Feasibility (capacity for pharmacist to implement) | 6 months
  Challenges regarding implementation for pharmacists from field notes and interviews
Feasibility (issues with TaperMD tool) | 6 months
  Communication between pharmacists and research team noting TaperMD issues from regular meetings.
Feasibility (missing data) | 6 months
  Nature and percentage of missing data.
Feasibility (variance of measures) | Baseline, 6 months
  The calculated range of scores for surveys (where applicable)
Feasibility (intervention implementation proportion) | 6 months
  Number of plans containing deprescribing actions divided by the total number of plans.

OTHER OUTCOMES:
Successful discontinuation | 6 months
  Mean difference in number of medications
Successful discontinuation or dose reduction | 6 months
  Composite variable calculate to represent mean number of medications stopped or dose reductions
Successful discontinuation or dose reduction (proportion) | 6 month
  Proportion of patients with successful discontinuation or dose reduction
Quality of life (EQ5D-5L) | Baseline, 6 months
  EuroQol five dimensions questionnaire (EQ5D-5L).
Quality of life (SF36v2) | Baseline, 6 months
  The Short Form (36) Health Survey (SF-36-V2).
Falls | Baseline, 6 months
  Total number of falls resulting in medication consultation or treatment recorded in hospital admission and primary care records, and by patient.
Fatigue | Baseline, 6 months
  Avlund Mob-T Scale
Pain severity and interference | Baseline, 6 months
  Brief Pain Inventory (Pain interference and Pain severity sub-scales)
Sleep | Baseline, 6 months
  15-D Scale (Sleep Question)
Treatment Burden | Baseline, 6 months
  Brief Treatment Burden Scale
Physical function capacity and ability (MANTY) | Baseline, 6 months
  Manty structured validated interview
Physical function capacity and ability (balance) | Baseline, 6 months
  Global Rating of Change (Balance).
Healthcare resource utilization (hospital admissions) | Baseline, 6 months
  Number of hospital admissions from administrative data and self-report; proportion of patients with at least one hospitalization.
Healthcare resource utilization (ED/urgent care visits) | Baseline, 6 months
  Number of emergency department and urgent care visits from administrative data and self-report.
Healthcare resource utilization (primary care visits) | Baseline, 6 months
  Number of primary care visits from administrative data
Changes in medication side effects and symptoms (adverse) | 1 week, 3 month, 6 month
  Patient self-report of appearance (new or worsening) of side effects associated with medications.
Changes in medication side effects and symptoms (positive) | 1 week, 3 month, 6 month
  Patient self-report of disappearance (improvement or disappearance) of side effects associated with medications.
Serious adverse events | Baseline, 6 months
  Any event that requires in-patient hospitalization or prolongation of existing hospitalization, causes congenital malformation, results in persistent or significant disability or incapacity, is life-threatening or results in death (Health Canada (2011) Guidance Document for Industry - Reporting Adverse Reactions to Marketed Health Products).
Implementation processes | Baseline, 3 months, 6 months
  NoMAD survey
Pharmacists/family physician 5 best/worst aspects of intervention | 6 months
  Open ended list
Pharmacists/family physician confidence in medication discontinuation | Baseline, 6 months
  5 point Likert scale single question developed for study
Pharmacists/family physician experiences with the deprescribing process | 6 months
  Semi-structured interviews; field notes
Patient experience with deprescribing process (interview) | 6 months
  Semi-structured interview
Satisfaction with intervention | 6 months
  5 point Likert scale single question developed for study
Satisfaction with care around medications | Baseline, 6 months
  5 point Likert scale single question developed for study

CONTACTS AND LOCATIONS:
Locations (1):
- Dr. Dee Mangin, Hamilton, Ontario, Canada

IPD SHARING:
Plan to Share IPD: Undecided